CLINICAL TRIAL: NCT02114866
Title: Quality of Handover to a Post Anaesthesia Care Unit in a Children's Hospital
Status: Completed | Type: Observational
Sponsor: University of Witten/Herdecke (Other)
Responsible Party: Principal Investigator, Florian Piekarski, Doctoral candidate, University of Witten/Herdecke
Other Study IDs: 110/2012
Record Dates: First submitted 2014-04-10; First posted 2014-04-15 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-04

CONDITIONS: Information Transfer During Postoperative Handovers

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Postoperative handovers to the post anaesthesia care unit (PACU) in adult anaesthesia are described as incomplete and unstructured, although their relevance for the patient safety is well known. It must be assumed that for children, this handover is at least comparable important.

With a self-developed checklist information transfer during postoperative handovers will be documented and subsequently compared with patient information in anaesthesia records.

ELIGIBILITY:
Inclusion Criteria:

* All patients transferred to the PACU after surgery

Exclusion Criteria:

* Age > 18 years

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population consists of patients (<18 years of age) at Children's Hospital Cologne, being admitted to the main postoperative care unit (PACU), after they underwent interventions within normal surgery hours
Sampling Method: Probability Sample
Enrollment: 441 (Actual)
Dates: Start 2012-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Quantity of Information Loss during Postoperative Handovers in the PACU | Three month

REFERENCES:
- [Derived] Piekarski F, Kaufmann J, Laschat M, Bohmer A, Engelhardt T, Wappler F. Quality of handover in a pediatric postanesthesia care unit. Paediatr Anaesth. 2015 Jul;25(7):746-52. doi: 10.1111/pan.12646. Epub 2015 Apr 2. PMID 25833388